CLINICAL TRIAL: NCT03609996
Title: A Retrospective Review of Patients With Proliferative Diabetic Retinopathy and Regression of PDR After Treatment With Ranibizumab
Brief Title: Retrospective Review of Proliferative Diabetic Retinopathy Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Elman Retina Group (Other)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29652
Record Dates: First submitted 2018-07-24; First posted 2018-08-01 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- PDR treated with Laser
  Interventions: Device: Panretinal Photocoagulation; Drug: Lucentis
- PDR treated with Lucentis
  Interventions: Device: Panretinal Photocoagulation; Drug: Lucentis

INTERVENTIONS:
Device: Panretinal Photocoagulation — Laser treatment for PDR
Drug: Lucentis — Intraviteral injection

SUMMARY:
The primary objective of the protocol is to determine if intravitreal ranibizumab alone decreases retinal neovascularization from Proliferative Diabetic Retinopathy (PDR) with deferred panretinal photocoagulation (PRP) and/or vitrectomy at one year after treatment with ranibizumab has been initiated.

DETAILED DESCRIPTION:
Current standard treatment for Proliferative Diabetic Retinopathy (PDR) is panretinal photocoagulation (PRP), but this treatment is inherently destructive and has several potential adverse effects on aspects of visual function, including constriction of peripheral visual fields and decreases in night vision, contrast sensitivity and color perception. Thus, therapeutic alternatives that might delay or obviate the need for PRP are desirable. It has been demonstrated that retinal neovascularization from PDR is highly responsive to anti-VEGF therapy, but it is unclear how long regression of retinal neovascularization is sustained after anti- VEGF therapy is halted in clinical practice.

It is possible that intravitreal ranibizumab treatment could prevent laser-associated vision loss by precluding the need for PRP as long as the eye continued to receive ranibizumab. Even if ranibizumab treatment was discontinued, it is possible that initial treatment with anti-VEGF therapy might improve visual outcomes substantially by delaying or preventing the need for PRP, and the infrequent frequency of administration of ranibizumab for DME (median 2 to 3 times in the second year of treatment) after the DME initially has resolved on anti-VEGF therapy suggests that monthly ranibizumab might not be needed to achieve control of PDR.

The Diabetic Retinopathy Clinical Research Network (DRCR network) is currently evaluating intravitreal ranibizumab treatment to see if can prevent laser-associated vision loss by precluding the need for PRP as long as the eye continued to receive ranibizumab. However, intravitreal injections carry the risk of serious complications. Ophthalmic complications include endophthalmitis in 2% of all injected patients cumulatively. Endophthalmitis is a vision threatening and can cause severe and permanent vision loss and even loss of the eye. Other complications include vitreous hemorrhage, retinal detachment, uveitis and glaucoma. This study will evaluate ranibizumab usage as the primary treatment for PDR in a busy private clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years Individuals <18 years old are not being included because PDR is so rare in this age group that the diagnosis of PDR may be questionable.
2. Diagnosis of diabetes mellitus (type 1 or type 2)

   Any one of the following will be considered to be sufficient evidence that diabetes is present:
   * Current regular use of insulin for the treatment of diabetes
   * Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes
   * Documented diabetes by ADA and/or WHO criteria (see Procedures Manual for definitions
3. Presence of PDR which the investigator has treated the study eye(s) with ranibizumab

Exclusion Criteria:

1. History of prior panretinal photocoagulation prior to initiating ranibizumab
2. Tractional retinal detachment involving the macula.

   * A tractional retinal detachment is not an exclusion if it is outside of the posterior pole (not threatening the macula)
3. History of vitrectomy prior to initiating ranibizumab
4. Treatment with Ranibizumab within six months of treatment regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 160 eyes that have been diagnosed with PDR that have been treated with ranibizumab will be looked at retrospectively.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical regression of neovascularization not requiring further treatment beyond RBZ | 2009-2018
  Clinical regression of neovascularization not requiring further treatment beyond RBZ

CONTACTS AND LOCATIONS:
Overall Officials: Michael Elman, Principal Investigator — Elman Retina Group, P.A.
Locations (1):
- Elman Retina Group, Baltimore, Maryland, United States